CLINICAL TRIAL: NCT06513884
Title: A Randomized Double-blinded Phase 2/3 Study of HB-202/HB-201 Alternating 2-Vector Therapy With Pembrolizumab Versus Pembrolizumab-Only for First Line HPV16+ High PD-L1 CPS Recurrent and/or Metastatic Oropharyngeal Squamous Cell Carcinoma
Brief Title: A Study of HB-202/HB-201 With Pembrolizumab in Patients With HPV16+ Recurrent/Metastatic Oropharyngeal Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the decision by the company not to pursue the development of HB-202 and HB-201 in this indication.
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-200-004
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-02

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma Recurrent
Keywords: head and neck cancer; squamous cell cancer; head and neck squamous cell carcinoma; HNSCC; oropharyngeal squamous cell carcinoma; human papillomavirus 16; HPV; programmed cell death 1 ligand 1; PD-L1; immune checkpoint inhibitor; immunotherapy; genetic vector; arenavirus
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HB-202/HB-201 alternating 2-vector therapy with pembrolizumab (Experimental): Intravenous injection of HB-202 followed by pembrolizumab alternating with HB-201 followed by pembrolizumab.
  Interventions: Drug: HB-202/HB-201 alternating 2-vector therapy; Drug: Pembrolizumab
- Matched placebo with pembrolizumab (Placebo Comparator): Intravenous injection of matched placebo for HB-202 followed by pembrolizumab alternating with matched placebo for HB-201 followed by pembrolizumab.
  Interventions: Drug: Placebo; Drug: Pembrolizumab

INTERVENTIONS:
Drug: HB-202/HB-201 alternating 2-vector therapy — Intravenous administration of HB-202 alternating with HB-201, with the first 2 treatment cycles administered every 3 weeks and then every 6 weeks from the third treatment cycle onwards.
  Other Names: HB-202 intravenous administration alternating with HB-201 intravenous administration; HB-201 & HB-202 two-vector therapy; TheraT® Vector(s) Expressing Human Papillomavirus 16 Positive (HPV16+) Specific Antigens
  Arms: HB-202/HB-201 alternating 2-vector therapy with pembrolizumab
Drug: Placebo — Intravenous administration of matched placebo for HB-202 alternating with matched placebo for HB-201, with the first 2 treatment cycles administered every 3 weeks and then every 6 weeks from the third treatment cycle onwards.
  Other Names: Matched placebo
  Arms: Matched placebo with pembrolizumab
Drug: Pembrolizumab — Intravenous administration of pembrolizumab, with the first 2 treatment cycles administered at a dosage of 200 mg every 3 weeks and then every 6 weeks from the third treatment cycle onwards administered at a dosage of 400 mg.
  Other Names: Keytruda®

SUMMARY:
This is a study of HB-202/HB-201 alternating 2-vector therapy with pembrolizumab (also known as Keytruda®) in people with human papillomavirus subtype 16 positive (HPV16+) head and neck cancer starting in the middle part of the throat, who have not yet received systemic treatment after their cancer spread (metastatic) and/or returned (recurrent) and who are eligible to receive pembrolizumab.

Doctors already use pembrolizumab therapy (with or without chemotherapy) to treat head and neck cancer. However, the treatment does not work well in most people with this type of cancer. HB-202/HB-201 alternating 2-vector therapy with pembrolizumab, which is designated to stimulate a stronger immune attack against HPV16+ tumors, was shown to be safe and suggested to work better than pembrolizumab-only in a small number of participants with HPV16+ head and neck cancer (see H-200-001, NCT04180215).

This trial studies HB-202/HB-201 alternating 2-vector therapy with pembrolizumab in a much larger number of participants from different countries to confirm its benefits for people with HPV16+ head and neck cancer that started in the middle part of the throat compared with pembrolizumab-only therapy. This trial studies whether administering HB-202/HB-201 alternating 2-vector therapy with pembrolizumab works better in more participants by shrinking their tumors and makes them live longer than pembrolizumab-only therapy.

Participants will receive the study treatments by injection into a vein every 3 weeks during the first 3 months and then every 6 weeks until up to about 2 years, which will be followed by a long observation period to continue looking at the safety and clinical benefits after the last dose of study treatment.

DETAILED DESCRIPTION:
This is a seamless adaptive Phase 2/3, randomized, double-blinded, placebo-controlled, multicenter trial of HB-202/HB-201 alternating 2-vector therapy with the approved drug pembrolizumab in participants with HPV16+ recurrent and/or metastatic oropharyngeal squamous cell carcinoma (OPSCC), whose tumor has a programmed cell death ligand-1 (PD-L1) combined positive score (CPS) greater than or equal to 20 in the first line setting. OPSCC is a type of head and neck squamous cell carcinoma (HNSCC) originating in the oropharyngeal region (tonsil, tongue base, soft palate, or uvula). The study will evaluate the long-term safety and the benefits on objective response rate, overall survival, and progression-free survival of HB-202/HB-201 alternating 2-vector therapy plus pembrolizumab compared with pembrolizumab-only therapy.

Pembrolizumab-only therapy or pembrolizumab plus chemotherapy are currently the first-line therapies used to treat people with recurrent and/or metastatic HNSCC (including HPV+ OPSCC). However, poor prognosis prevails despite pembrolizumab therapy with or without chemotherapy (including patients with PD-L1 CPS greater or equal to 20), where only a minority of patients respond.

HB-202 and HB-201 are genetically engineered, replicating vectors based on the arenaviruses Pichinde virus and lymphocytic choriomeningitis virus, respectively. The HB-202 and HB-201 vectors have been engineered to deliver specific non-oncogenic antigens derived from HPV16, which enables the vectors to stimulate a strong and specific immune response against HPV16+ tumor cells. Pembrolizumab on the other hand is a potent checkpoint inhibitor, which binds to immune cell surface receptors to relieve the typical inhibition of immune surveillance of tumors. In an early phase trial (H-200-001, NCT04180215), HB-202/HB-201 alternating 2-vector therapy with pembrolizumab has shown favorable safety and preliminary anti-tumor activity with an objective response rate higher than previously reported with pembrolizumab-only therapy in participants with HPV16+ OPSCC.

HB-202/HB-201 alternating 2-vector therapy or matched placebo will be administered in treatment cycles. A treatment cycle is defined as one administration of HB-202 plus the post-dose period followed by one administration of HB-201 plus the post-dose period until the next dose. In the first 2 treatment cycles, the HB-202/HB-201 or matched placebo treatment is administered with 200 mg pembrolizumab every 3 weeks. The HB-202/HB-201 or matched placebo treatment is administered with 400 mg pembrolizumab every 6 weeks from the third treatment cycle onwards. Adverse events (AEs) will be monitored for up to 30 days and serious AEs for up to 90 days after the last dose of study treatment. There will be long-term follow-up every 3 months after the last administration of study treatment for all participants until the participant's death, the participant is lost to follow-up or withdraws consent to follow-up, last study-related phone call or visit, or study termination, whichever occurs first.

Participants will be randomized to receive either HB-202/HB-201 alternating 2-vector therapy followed by pembrolizumab or matched placebo (i.e., matched to the respective viral vector) followed by pembrolizumab.

Up to 150 Investigators and study sites in North America, Europe, and other regions of the world are expected to enroll participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years of age.
* Confirmed recurrent and/or metastatic OPSCC that is considered incurable by local therapies.
* Must not have had prior systemic anticancer therapy, including investigational therapy and non-palliative radiotherapy, administered in the recurrent and/or metastatic setting.
* Confirmed HPV16+ AND PD-L1+ (with a CPS greater or equal to 20) tumor, based on tumor specimen, core, or excisional biopsy samples from a tumor lesion not previously irradiated.
* Must have measurable disease based on RECIST version 1.1 as determined by BICR.
* Eastern Cooperative Oncology Group performance status must be 0 to 1.
* Adequate organ function should be confirmed within 10 days prior to the first dose of study treatment.

Exclusion Criteria:

* Has progressive disease within 6 months of completion of curatively intended systemic treatment (including checkpoint inhibitors) for locoregionally advanced OPSCC.
* Life expectancy of less than 3 months and/or rapidly progressing disease, high burden of visceral metastatic disease, or significant tumor burden in anatomically critical areas (e.g., causing significant biliary or respiratory obstruction) who may benefit from a chemotherapy-based treatment regimen.
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the trial or interfere with the participant's participation for the full duration of the trial, or such that it is not in the best interest of the patient to participate, in the opinion of the treating Investigator. This includes active cardiovascular disease within 6 months before study entry.
* Is pregnant or breastfeeding or expecting to conceive or father children starting with the screening visit through a minimum of 2 months after the last dose of trial treatment.
* Was discontinued due to a Grade 3 or 4 immune-related AE after receiving prior therapy with a checkpoint inhibitor agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Received systemic steroids at a dose of >10 mg/day (prednisone equivalent) for <30 days within 14 days or for ≥30 days within 28 days of the first dose of study treatment.
* Received live, or live-attenuated vaccine within 30 days of the planned first dose of treatment or anticipates that such a vaccine will be required during the study.
* Participating in or has participated in a study of an investigational agent, or has used an investigational device treatment, within 4 weeks before the first dose of study treatment.
* Has had an allogeneic tissue/solid organ transplant.
* Has known immunodeficiency OR is receiving long-term systemic steroid therapy or any other form of immunosuppressive therapy within 28 days before the first dose of study treatment.
* Known additional malignancy within 2 years before the first dose of study treatment.
* Known CNS metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (Grade 3 and/or 4) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* History or current evidence of (non-infectious) pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Known history of acquired immunodeficiency syndrome (AIDS). Testing for human immunodeficiency virus (HIV) is not mandatory.
* Known history of hepatitis B virus (defined as hepatitis B surface antigen reactive) or known active hepatitis C virus infection (defined as hepatitis C virus ribonucleic acid [RNA] is detected [qualitative]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate - Blinded independent central review (BICR) | Up to 7.5 years after first dose of study treatment
  Objective response rate (ORR) defined as the proportion of participants with a confirmed best overall response of complete response or partial response, as assessed by BICR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival | Up to 7.5 years after first dose of study treatment
  Overall survival defined as the time from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-free survival - BICR | Up to 7.5 years after first dose of study treatment
  Progression-free survival (PFS) defined as the time from the date of randomization to the date of progressive disease, as assessed by BICR based on RECIST version 1.1, or to the date of death from any cause, whichever occurs first.
Duration of response - BICR | Up to 7.5 years after first dose of study treatment
  Duration of response (DOR) defined as the time from the date of the first objective response (complete or partial response) to the date of progressive disease as assessed by BICR based on RECIST version 1.1, or to the date of death from any cause, whichever occurs first.
Disease control rate - BICR | Up to 7.5 years after first dose of study treatment
  Disease control rate (DCR) defined as the proportion of participants with a confirmed best overall response of complete response, partial response, or stable disease as assessed by BICR based on RECIST version 1.1.
Progression-free survival on next-line therapy | Up to 7.5 years after first dose of study treatment
  Progression-free survival on next-line therapy defined as the time from the date of randomization to the Investigator-reported date of progression on next-line therapy, or to the date of death from any cause, whichever occurs first.
Objective response rate - Investigator | Up to 7.5 years after first dose of study treatment
  ORR defined as the proportion of participants with a confirmed best overall response of complete response or partial response, as assessed by the Investigator based on RECIST version 1.1 and immune RECIST (iRECIST).
Progression-free survival - Investigator | Up to 7.5 years after first dose of study treatment
  PFS defined as the time from the date of randomization to the date of progressive disease, as assessed by the Investigator based on RECIST version 1.1 and iRECIST, or to the date of death from any cause, whichever occurs first.
Duration of response - Investigator | Up to 7.5 years after first dose of study treatment
  DOR defined as the time from the date of the first objective response (complete or partial response) to the date of progressive disease as assessed by the Investigator based on RECIST version 1.1 and iRECIST, or to the date of death from any cause, whichever occurs first.
Disease control rate - Investigator | Up to 7.5 years after first dose of study treatment
  DCR defined as the proportion of participants with a confirmed best overall response of complete response, partial response, or stable disease as assessed by the Investigator based on RECIST version 1.1 and iRECIST.
Proportion of participants with AEs - overall | Up to 7.5 years after first dose of study treatment
  Overall occurrence of AEs by relationship to study treatment, type, grade, and seriousness.
Adjusted on-study year rate of AEs | Up to 7.5 years after first dose of study treatment
  Adjusted on-study yearly rate of AEs by relationship to study treatment, type, grade, and seriousness.
Proportion of participants with laboratory abnormality - overall | Up to 2 years after first dose of study treatment
  Overall occurrence of laboratory abnormality by laboratory test.
Adjusted on-study yearly rate of laboratory abnormality | Up to 2 years after first dose of study treatment
  Adjusted on-study yearly rate of laboratory abnormality by laboratory test.
Participant-reported health-related quality of life - European Quality of Life scale EQ-5D-3L | Up to 7.5 years after first dose of study treatment
  European Quality of Life 5 Dimensions 3 Level (EQ-5D-3L) score by dimension and item.
Participant-reported health-related quality of life - EORTC QLQ-C30 | Up to 7.5 years after first dose of study treatment
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) score by scale and item.
Participant-reported health-related quality of life - EORTC QLQ-H&N35 | Up to 7.5 years after first dose of study treatment
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck Cancer module 35 (EORTC QLQ-H&N35) score by scale and item.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, Study Director — Hookipa Biotech GmbH

IPD SHARING:
Plan to Share IPD: No